Date: 04.05.2020 Version: 3

## **STATISTICAL ANALYSIS PLAN**

Study name: Evaluation Of The Effectiveness And Safety Of Adding Ivermectin to

Treatment in Severe COVID-19 Patients

**Study protocol cod:** IVMC\_03

**Ethics committee approval number and date:** 139/03.04.2020

Coordinator researcher: Prof. Dr. Nurullah OKUMUŞ

## STATISTICAL ANALYSIS PLAN

Convenience Sampling method will be used in the study. Unilateral blinding will be made in determining which of the study and control groups participating patients will be included in the study, those with an odd number will be included in the study group, and those with an even number will be included in the control group.

In determining the sample size, it was planned to include 30 individuals in each group based on the number of available kits. In this case, the values of 0.05 for Type I Error Rate, 0.67 for Effect Size and 0.80 for Power were reached.

The Chi-Square test will be used in the evaluation of categorical data, the Wilcoxon test for in-group comparisons, and the Mann-Whitney U test for intergroup comparisons. For statistical significance, the value of p=0.05 will be taken into account and the analyzes will be carried out in the SPSS 20.0 package program.